CLINICAL TRIAL: NCT01787331
Title: Hedgehog Inhibition as a Non-Castrating Approach to Hormone Sensitive Prostate Cancer: A Phase II Study of Itraconazole in Biochemical Relapse
Brief Title: Itraconazole in Treating Patients With Biochemically Relapsed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 125513; NCI-2013-02375 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage I Prostate Adenocarcinoma AJCC v7; Stage II Prostate Adenocarcinoma AJCC v7; Stage III Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (itraconazole) (Experimental): Patients receive twice/day 300mg itraconazole (oral)
  Interventions: Drug: Itraconazole; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Itraconazole — Given PO
  Other Names: Lozanoc; Oriconazole; R 51,211; Sporanox
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well itraconazole works in treating patients with biochemically relapsed prostate cancer. Itraconazole may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the proportion of patients who achieve a >= 50% decline in serum prostate-specific antigen (PSA) after 12 weeks of protocol therapy with itraconazole dosed at 300 mg orally (PO) twice daily (BID) is superior to a historical control based upon the observed PSA response proportion in prior studies of non-castrating systemic therapy in men with biochemically relapsed hormone sensitive prostate cancer.

SECONDARY OBJECTIVES:

I. To determine the median time to PSA progression from the start of protocol therapy with itraconazole among men with biochemically relapsed prostate cancer.

II. To determine the median time to clinical progression measured from the start of protocol therapy with itraconazole among men with biochemically relapsed prostate cancer.

III. To determine the median metastasis-free survival measured from the start of protocol therapy in patients treated with itraconazole for biochemically relapsed prostate cancer.

IV. To determine the mean percent change from baseline after 12 weeks of protocol therapy compared with pre-treatment in PSA doubling time.

V. To characterize the safety profile of itraconazole in the biochemically relapsed hormone sensitive prostate cancer population, as graded by Common Toxicity Criteria (CTCAE) version 4.03. All adverse events will be tabulated by grade according to the worst grade experienced.

VI. To determine the mean steady-state itraconazole and hydroxy-itraconazole serum levels after 4 weeks of therapy with itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate
* Biochemically relapsed disease with a rising PSA on at least two successive measurements at least two weeks apart after prior definitive local therapy (radical prostatectomy, external beam radiation, or brachytherapy) or combination of radical prostatectomy and radiotherapy (RT) with curative intent; if the confirmatory PSA value is less than the screening PSA value, then an additional test for rising PSA will be required to documents progression
* Prior primary or salvage radiation or not a candidate for salvage radiation due to patient preference or clinical assessment based upon disease characteristics and/or patient co-morbidities
* Minimum PSA:

  * If no prior androgen deprivation therapy (ADT) for biochemical relapse:

    * 1.0 ng/mL if prior radical prostatectomy with or without adjuvant/salvage radiation therapy, confirmed by repeat measurement at least 2 weeks later, or
    * Nadir + 2 ng/mL if prior RT alone without prior radical prostatectomy, confirmed by repeat measurement at least 2 weeks later
  * If prior ADT for biochemical relapse:

    * 4.0 ng/mL or > 2 ng/mL above nadir on prior cycle of ADT, whichever is higher, confirmed by repeat measurement at least 2 weeks later
* No evidence of metastatic disease on imaging by whole body bone scan (technetium-99 or sodium fluoride [Na-F] positron emission tomography [PET] bone scan) and cross-sectional imaging of the abdomen/pelvis (computed tomography [CT] or magnetic resonance imaging [MRI]) within 6 weeks of day 1 of protocol therapy
* Prior androgen deprivation therapy (ADT) with luteinizing hormone-releasing hormone (LHRH) agonist and/or antagonist allowed for either (neo)adjuvant treatment with local therapy or for biochemical relapse
* Last effective dose of LHRH agonist/antagonist ?expired? > 3 months prior to study entry; for example, a patient receiving LHRH agonist injection every 3 months would be eligible provided their last injection was > 6 months prior to day 1 of protocol therapy; a patient receiving LHRH agonist injections every 4 months will be eligible provided last injection was > 7 months prior to day 1 of protocol therapy
* Serum testosterone level:

  * If no prior androgen deprivation therapy:

    * A single measurement greater than 150 ng/dL within 3 months of day 1 of protocol therapy
  * If prior androgen deprivation therapy (either in adjuvant or biochemical relapse setting):

    * The two most recent measurements of serum testosterone prior to day 1 of protocol therapy must fulfill the following criteria:

      * Both measurements are greater than 150 ng/dL
      * The two measurements are spaced at least 14 days apart
      * Both must be measured within 3 months of day 1 of protocol therapy
      * There must not be an increase of > 50 ng/dL between these two successive measurements
* PSA doubling time (PSADT) =< 15 months, calculated based upon all serum PSA measurements obtained within 3 months prior to day 1 of protocol therapy, with a minimum of three PSA measurements spaced at least 14 days apart ; PSA values obtained when serum testosterone was known to be less than 150 ng/dL, prior to local therapy, or within three months of last dose of LHRH agonist/antagonist or antiandrogen will be excluded from the calculation of the PSADT
* Total bilirubin less than 1.5 times upper limit of normal (ULN), or less than 3 times ULN at study entry in a patient with documented Gilbert?s disease
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels less than 1.5 times ULN at study entry
* Serum potassium greater than 3.5 mmol/L without oral supplementation
* No history of uncontrolled hypertension (blood pressure > 160/100 mm Hg despite anti-hypertensive medication)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Estimated life expectancy greater than 5 years
* Ability to sign written informed consent
* Ability to swallow study drug whole as a capsule
* Primary prostate cancer tissue available for analysis is not required for inclusion onto this study but is strongly encouraged
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last study drug administration

Exclusion Criteria:

* Castrate-resistant disease, as evidenced by either:

  * Rising PSA on 2 consecutive measurements at least 2 weeks apart with concurrent documented serum testosterone < 50 ng/dL at the time of PSA measurement, or
  * Rising PSA on 2 consecutive measurements at least 2 weeks apart measured within 3 months after last LHRH agonist/antagonist injection
* Prior bilateral orchiectomy
* Congestive heart failure of New York Heart Association (NYHA) class III or higher severity at study entry
* History of chronic active hepatitis
* Grade 2 or higher peripheral neuropathy at the time of study entry
* Use of 5-alpha reductase antagonist (i.e. finasteride, dutasteride) or antiandrogen (i.e. flutamide, bicalutamide) within 6 weeks of day 1 of protocol therapy
* Use of systemic steroids at an equivalent dose of prednisone 5 mg/day or higher within 6 weeks of day 1 of protocol therapy
* Use of medications or herbal supplements which are known to potentially lower serum PSA within 6 weeks of day 1 of protocol therapy
* Use of other medications that may potentially interact with itraconazole within 1 week of study entry
* Use of other investigational agents within 6 weeks of day 1 of protocol therapy
* Prior pathology consistent with small cell carcinoma or prostate cancer with predominantly neuroendocrine differentiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mina Lee, Haemin Hong, Won Kim, Terence W. Friedlander, Lawrence Fong, Amy M. Lin, Eric Jay Small, Mallika Sachdev Dhawan, Xiao X. Wei, Tammy J. Rodvelt, Brigid Miralda, Charles J. Ryan, and Rahul Raj Aggarwal.A phase II study of itraconazole in biochemically recurrent prostate cancer. Journal of Clinical Oncology 2018 36:6_suppl, 362-362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Itraconazole)
Started | 21
Completed | 19
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 21
Age, Customized [Number; unit: participants]
  40-49 Years | 1
  50-59 Years | 1
  60-69 Years | 10
  70-79 Years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Years since diagnosis of prostate cancer [Mean (Full Range); unit: years] | 7.83 [0.63 to 18.01]
Gleason Grade at Time of Diagnosis [Count of Participants; unit: Participants] — Gleason grade is determined at the time of diagnosis based on pathology review of prostate cancer biopsy or surgical specimen. A higher Gleason grade (> 7) is associated with a higher chance for disease recurrence and shorter long-term survival.
  Participants
    Gleason grade ≤ 7 (low/intermediate grade) | 14
    Gleason grade > 7 (high grade) | 7
Time interval from biochemical relapse to study entry [Mean (Full Range); unit: years] | 4.01 [0.13 to 16.44]
PSA doubling time at the time of study entry [Mean (Full Range); unit: months] | 5.72 [1.16 to 13.05]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve a Greater Than or Equal to 50% Decline in Serum Prostate Specific Antigen (PSA)
Description: The number of patients with biochemically relapsed disease after prior definitive local therapy who achieve a ≥ 50% decline from baseline in serum PSA after 12 weeks of therapy with itraconazole, confirmed by repeat measurement at least 2 weeks later.
Time Frame: At 12 weeks after start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 19
Participants | 1

2. Secondary Outcome: Mean Percent Change in PSA Doubling Time
Description: The mean percent change in PSA doubling time from pre-treatment to after 12 weeks of protocol therapy
Time Frame: Up to 12 weeks
Measure: Mean (Full Range); unit: Percent change in PSA doubling time
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 19
Percent change in PSA doubling time | -0.64 [-59.96 to 71.38]

3. Secondary Outcome: Median Time to PSA Progression
Description: PSA progression defined as: 1. If no PSA decline is observed on therapy, PSA progression will be defined as an increase in serum PSA > 50% above the baseline PSA, and an absolute increase of > 2 ng/mL above baseline, confirmed by repeat measurement at least 2 weeks later. 2. If PSA declines on therapy, PSA progression will be defined as an increase in serum PSA > 50% above the nadir PSA on therapy, and an absolute increase > 2 ng/mL above the nadir, confirmed by repeat measurement at least 2 weeks later. The probability distribution of the time to PSA progression will be estimated using the Kaplan-Meier product limit method measured from the start of protocol therapy. The results will be summarized by the estimated median with 95% confidence intervals.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 19
months | 4.68 [2.0 to 21.7]

4. Secondary Outcome: Median Time to Clinical Progression
Description: Clinical progression will be defined as the first occurrence of either the development of metastases or initiation of non-protocol therapy, and will exclude PSA-only progression.
  The probability distribution of the time to clinical progression will be estimated using the Kaplan-Meier product limit method measured from the time of start of protocol therapy. The results will be summarized by the estimated median with 95% confidence intervals.
Time Frame: Up to 2 years
Population: Only 1 patient displayed clinical progression
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 1
months | 21.7 [21.7 to 21.7]

5. Secondary Outcome: Median Metastasis-free Survival
Description: The probability distribution of the time to first metastasis will be estimated using the Kaplan-Meier product limit method measured from the time of start of protocol therapy. The results will be summarized by the estimated median with 95% confidence intervals.
Time Frame: Up to 2 years
Population: Data not collected
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants With Treatment-related, Adverse Changes in Vital Signs
Description: All patients who receive at least one dose of study drug will be analyzed for safety endpoints. All adverse events will be graded and classified according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 4. Percentage of patients with grade 1 or higher, treatment-related adverse events based on the following vital sign assessments will be reported: blood pressure, pulse, respiration rate and temperature.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 21
percentage of participants
  Blood Pressure | 14.3
  Weight | 0
  Pulse | 0
  Respiration Rate | 0
  Temperature | 0

7. Secondary Outcome: Percentage of Participants With Treatment-related, Clinical Laboratory Adverse Events
Description: All patients who receive at least one dose of study drug will be analyzed for safety endpoints. All adverse events will be graded and classified according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 4.. Percentage of patients with grade 1 or higher, treatment-related adverse events based on the following labs will be reported: potassium, sodium, alkaline phosphatase, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), Hematocrit, Hemoglobin, platelets, white blood cells, atypical lymphs, basophils, eosinophils, monocytes, neutrophils, blood urea nitrogen, and creatinine.
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 21
percentage of participants
  Potassium | 9.52
  Alanine aminotransferase | 4.76
  Sodium | 0
  Alkaline phosphatase | 0
  Total bilirubin | 0
  Aspartate aminotransferase | 0
  Hematocrit | 0
  Hemoglobin | 0
  Platelets | 0
  White blood cells | 0
  Atypical lymphs | 0
  Basophils | 0
  Eosinophils | 0
  Monocytes | 0
  Neutrophils | 0
  Blood urea nitrogen | 0
  Creatinine | 0

8. Secondary Outcome: Mean Steady-state Trough Level of Serum Itraconazole
Description: Descriptive statistics including the mean, standard deviation, and range of steady-state trough serum levels of itraconazole and its active metabolite hydroxy-itraconazole will be determined.
Time Frame: Up to 4 weeks
Population: No data collected
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Steady-state Trough Level of Hydroxy-itraconazole
Description: as for outcome 8
Time Frame: Up to 4 weeks
Population: No data collected
Arm/Group | Treatment (Itraconazole)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: All patients who received at least one dose of study drug were analyzed for adverse events
Arm/Group | Treatment (Itraconazole)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Itraconazole) (N=21)
Atrial flutter (Cardiac disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Investigations - Other, specify (Investigations) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Itraconazole) (N=21)
Edema limbs (General disorders) | 12
Fatigue (General disorders) | 9
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 6
Hot flashes (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Upper respiratory infection (Infections and infestations) | 5
Rhinitis infective (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
No evaluable data was collected from validated assay. Long term, metastatic disease status data was also not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT01787331/Prot_SAP_000.pdf